CLINICAL TRIAL: NCT00765258
Title: Utility of CT Fluoroscopy Guidance During Percutaneous Sacroplasty With Quality of Life Assessment
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Winthrop University Hospital (Other)
Responsible Party: Principal Investigator, Sean Tutton, MD, Principal Investigator, Medical College of Wisconsin
Other Study IDs: PRO00008209
Record Dates: First submitted 2008-09-30; First posted 2008-10-02 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2013-08

CONDITIONS: Sacro-iliac Insufficiency Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To examine, through retrospective and prospective chart review, the difference in pain and mobility, pre and post treatment, as assessed by the patient's completion of the VAS pain scale and Roland Morris Disability Questionnaire (RMDQ).

CT fluoroscopy guidance during percutaneous sacroplasty is an effective treatment for sacro-iliac insufficiency fractures resulting in rapid reduction of pain and improved mobility in patients. This can be effectively assessed using the VAS pain scale and RMDQ both pre and post procedure.

DETAILED DESCRIPTION:
The purpose of the study is to report the use of CT fluoroscopy guidance during the performance of percutaneous sacroplasty. In addition, clinical results will be reported with the Roland Morris Disability Questionnaire(RMDQ)pre and post procedure, demonstrating the utility of the RMDQ in assessing improvement in patients pain, mobility and ability to perform activities of daily living.

ELIGIBILITY:
Inclusion Criteria:

* greater than 18 years of age and treated with or about to be treated with percutaneous CT fluoro-guided sacroplasty, regardless of gender or ethnicity.

Exclusion Criteria:

* less than 18 years old
* pregnancy
* inability to complete forms and surveys

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient's with pain and decreased mobility as a result of sacro-iliac insufficiency fracture(s).
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2008-01; Primary Completion 2012-05 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Reduction of pain and improved mobility in patients post percutaneous sacroplasty effectively assessed using the VAS pain scale and RMDQ both pre and post procedure. | 2008-2012
  The average pre-treatment VAS score was significantly improved after sacroplasty in patients with sacral insufficiency fractures.

CONTACTS AND LOCATIONS:
Overall Officials: Sean M Tutton, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin / Froedtert Hospital, Milwaukee, Wisconsin, United States